CLINICAL TRIAL: NCT01612585
Title: A Registry Study on Safety Surveillance of Dengzhanxixin (a Chinese Medicine Injection) Used in China
Brief Title: Safety Study of Dengzhanxixin (a Chinese Medicine Injection) Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-Ⅴ; RSCMI-Ⅴ
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Ischemic Stroke; Coronary Heart Disease
MeSH Terms: conditions — Ischemic Stroke; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in October 2011.

It was funded by China major scientific and technological specialized project for 'significant new formulation of new drugs'.

Dengzhanxixin is kind of Chinese Medicine injection used for treating Ischemic Stroke and coronary heart disease in many Chinese hospitals.

The purpose of this study is to determine adverse drug events or adverse drug reaction in large sample size 30,000 patients.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China. However safety problems rose in recent years. There could be many uncertain factors influence Chinese Medicine Injection in clinical practice.

Safety surveillance on Chinese Medicine injection is an important problem that needs to be sorted out through large sample observational study.

A registry study for Kudiezi injection safety surveillance with 30000 patients will be conducted from April.2012 to December.2014.

Eligibility criteria Patients who will use Dengzhanxixin injection in selected hospitals

Data will be collected in three aspects by three different forms as following:

Form A (green): demographic information ；Form B (pink): adverse drug events/reaction； Form C (white): extracted information from hospital information system and laboratory information system Form

ELIGIBILITY:
Inclusion Criteria:

* Patients using Dengzhanxixin injection from 2012 to 2014

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 30000. Patients using Kudiezi injection from 2012 to 2014 in more than 30 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of Dengzhanxixin's ADRs and identify factors that contributed to the occurrence of the adverse reaction. | The registry procedure will last 3 years only for patients using Dengzhanxixin
  All patients will be measured and assessed at the time Dengzhanxixin is administered to them until they discharge. Patients using Dengzhanxixin will be registered on a registration form including disease background, Dengzhanxixin's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Dengzhanxixin.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences